CLINICAL TRIAL: NCT05275699
Title: Analyse of Diagnosis Value of Keloid on 68Ga- FAPI-04 PET-CT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-FAPI-KELOID
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-02

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-04 PET/CT (Experimental): All patients diagnosed with keloid underwent 68Ga-FAPI PET/CT.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 18.5-22.2MBq (0.5-0.6 mCi)/Kg 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of keloid by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
Keloid scars are common benign fibroproliferative reticular dermal lesions. Fibroblasts are considered to be the key cellular mediators of fibrogenesis in keloid scars. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may provide evidence for diagnosis and evaluate the effectiveness of treatment.

DETAILED DESCRIPTION:
Keloid scars are common benign fibroproliferative reticular dermal lesions with unknown etiology and ill-defined management with a high rate of recurrence post-surgery. The progression of keloids is characterized by increased deposition of extracellular matrix proteins, invasion of the surrounding healthy skin, and inflammation.

Fibroblast activation protein alpha (FAP-a) and dipeptidyl peptidase IV(DPPIV) are proteases located at the plasma membrane promoting cell invasiveness and tumor growth and have been previously associated with keloid scars. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment, and follow-up of keloid.

This study aims to explore whether FAP plays a role in the mechanisms of scar tissue progression, as well as the diagnostic efficacy of these two imaging agents, and to be able to evaluate relevant treatments for personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed pulmonary fibrosis patients;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for Lung fibrosis in comparison with 68Ga-RGD PET/CT

SECONDARY OUTCOMES:
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
therapy response | through study completion, an average of 1 year
  Change of 68Ga-FAPI PET/CT SUVmax after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang J, Yu N, Wang G, Wang R, Li L, Jiang Y, Sui H, Sun Y, Li Z, Long X, Zhu Z. 68 Ga-FAPI-04 PET/CT in Assessment of Fibroblast Activation in Keloids : A Prospective Pilot Study. Clin Nucl Med. 2024 Jan 1;49(1):16-22. doi: 10.1097/RLU.0000000000004913. Epub 2023 Nov 24. PMID 38015039